CLINICAL TRIAL: NCT03199027
Title: Timing of Referral to Adherence Clubs for Antiretroviral Therapy - a Randomised Controlled Trial
Brief Title: Timing of Referral to Adherence Clubs for Antiretroviral Therapy
Acronym: TRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Professor Landon Myer, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 764/2016
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Hiv
Keywords: Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-based Care (No Intervention): Clinic-based care is the current Standard-of-Care whereby newly initiated ART patients attend the ART clinic.
- Adherence Club Care (Experimental): Adherence club care involves referral to community-based ART services in the form of Adherence clubs, which are led by community health workers and supported by ART clinic nurses.
  Interventions: Other: Adherence Club

INTERVENTIONS:
Other: Adherence Club — Participants will be referred to an Adherence Club at 4 months post-ART initiation. Adherence club visits occur 2-4 monthly at a community hall near the Community Health Centre (CHC). At routine visits, which last 1-2 hours, community health workers provide health education, weigh patients, ask about symptoms and dispense pre-packed ART. Symptomatic patients are sent back to the ART clinic for clinician assessment. An assigned nurse takes blood tests annually at each club, and then returns on the subsequent visit to perform a clinical assessment and check the results. Patients requiring more follow-up or with high viral loads are referred back to the ART clinic at the CHC by the nurse.
  Arms: Adherence Club Care

SUMMARY:
Following the announcement of the global "90-90-90" strategy, there is a huge need in South Africa for effective well-developed scaled-up models of ART (anti-retroviral therapy) delivery that aim to improve patient adherence and viral suppression. The ART adherence club is one such model of service delivery. The investigators are conducting a pragmatic randomised control trial to compare virological outcomes 12 months post-ART initiation between arms: individuals referred to the Adherence club at 4 months post-ART initiation (early referral) and individuals referred to the Adherence club at 12 months post-ART initiation (delayed referral). Individuals with delayed Adherence club referral will continue to attend the ART clinic as per the Standard-of-Care.

DETAILED DESCRIPTION:
Following on from the huge need for scaled-up models of ART (anti-retroviral therapy) delivery to improve patient adherence and viral suppression, the ART adherence club model was piloted from 2007 with the aim of assessing whether this group-based, lay-counsellor led service, with an emphasis on social support and adherence, could help address retention in care and viral suppression. Since the initial pilots, the club model has been scaled up rapidly with more than 400 clubs meeting in the Cape Town metro. As this model is being scaled-up and implemented rapidly, there is an urgent necessity to further assess its effectiveness.

Whilst adherence clubs have been shown to be locally implementable, popular (with buy-in by clinic staff and patients) and cost-effective, and whilst community-based interventions have been shown to improve retention, evidence of local adherence club effectiveness in improving viral suppression and retention has only been observationally obtained. This observational evidence is highly subject to selection bias.

This trial aims to address this by using a randomised controlled trial design with two arms - ART patients receiving care in clinic as per the Standard-of-Care (this arm will have delayed referral to Adherence clubs at 12 months post-initiation) and ART patients receiving care in Adherence clubs (this arm will have early referral to Adherence clubs at 4 months post-initiation). By doing this the investigators hope to generate robust evidence regarding both the effectiveness of clubs and the optimal timing of club referral.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection with ART initiation 4 months ago
* Suppressed viral load at 4 months post-initiation (<400 copies/ml)
* All other month 4 blood results within normal limits
* Willingness to be randomised and return for study measurement visits
* Able to willing to attend service visits at either the clinic or a club
* Able to provide informed consent for research

Exclusion Criteria:

* Intention to relocate out of Cape Town permanently during the study period
* Any medical, psychiatric or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study
* Pregnant
* Current co-morbidity requiring additional health care, either acutely eg tuberculosis or chronically eg hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-10-06 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Viral suppression | Up to 12 months post-ART initiation
  Viral load <400 copies/ml with secondary analyses at other thresholds

SECONDARY OUTCOMES:
Retention in care | Up to 12 months post-ART initiation
  Numbers of missed visits and loss-to-follow up
Physical and Mental Health | Up to 12 months post-ART initiation
  As captured in the study visit questionnaires
Acceptability of the ART service | Up to 12 months post-ART initiation
  As captured in the study visit questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MBChB PhD, Principal Investigator — University of Cape Town
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luque-Fernandez MA, Van Cutsem G, Goemaere E, Hilderbrand K, Schomaker M, Mantangana N, Mathee S, Dubula V, Ford N, Hernan MA, Boulle A. Effectiveness of patient adherence groups as a model of care for stable patients on antiretroviral therapy in Khayelitsha, Cape Town, South Africa. PLoS One. 2013;8(2):e56088. doi: 10.1371/journal.pone.0056088. Epub 2013 Feb 13. PMID 23418518
- [Background] Grimsrud A, Sharp J, Kalombo C, Bekker LG, Myer L. Implementation of community-based adherence clubs for stable antiretroviral therapy patients in Cape Town, South Africa. J Int AIDS Soc. 2015 May 27;18(1):19984. doi: 10.7448/IAS.18.1.19984. eCollection 2015. PMID 26022654
- [Background] Grimsrud A, Lesosky M, Kalombo C, Bekker LG, Myer L. Implementation and Operational Research: Community-Based Adherence Clubs for the Management of Stable Antiretroviral Therapy Patients in Cape Town, South Africa: A Cohort Study. J Acquir Immune Defic Syndr. 2016 Jan 1;71(1):e16-23. doi: 10.1097/QAI.0000000000000863. PMID 26473798
- [Background] Takuva S, Brown AE, Pillay Y, Delpech V, Puren AJ. The continuum of HIV care in South Africa: implications for achieving the second and third UNAIDS 90-90-90 targets. AIDS. 2017 Feb 20;31(4):545-552. doi: 10.1097/QAD.0000000000001340. PMID 28121668